CLINICAL TRIAL: NCT02109744
Title: A Phase I/II Study of Decitabine in Combination With Sequential Rapamycin or Ribavirin in High Risk AML Patients
Brief Title: Study of Decitabine in Combination With Sequential Rapamycin or Ribavirin in High Risk AML Patients
Acronym: AML
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jane Liesveld, Principal INvestigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 48721; ULEU13049 (Other: University of Rochester)
Record Dates: First submitted 2013-10-14; First posted 2014-04-10 (Estimated); Results first posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decitabine followed by rapamycin (Experimental): Decitabine 20 mg/M2/day will be given as an IV infusion daily for 10 consecutive days starting on day 1 of cycle 1; in subsequent cycles, decitabine will be given for five days (days 1-5). Rapamycin 6mg (loading dose) will be administered on day 6; thereafter 2 mg/day on days 11-22 in cycle 1 and on days 6-22 in subsequent cycles. (Arm A: for patients with non-morphologic M4/M5 subtypes).
  Interventions: Drug: Decitabine
- Decitabine followed by ribavirin (Experimental): Decitabine 20 mg/M2/day will be given as an IV infusion daily for 10 consecutive days starting on day 1 of cycle 1; in subsequent cycles, decitabine will be given for five days (days 1-5). Ribavirin will be dosed from day 11-day 28 beginning with dose level 1 (1000mg orally twice daily). Number of patients with Dose Limiting Toxicities (DLT) at a given dose level is 0 of out of 3: enter 3 patients at the next dose level (dose Level 2- 1200mg orally twice daily; and then dose Level 3-1400 mg orally twice daily).(Arm B: For patients with morphologic M4/M5 subtypes).
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine
  Other Names: Dacogen; 5-aza-2'-deoxycytidine

SUMMARY:
To evaluate the response to chemotherapy with the drug decitabine combined with rapamycin in the treatment of relapsed or refractory acute myeloid leukemia in patients of all ages, and in the treatment of newly diagnosed leukemia in those who are older than 65 when diagnosed.

DETAILED DESCRIPTION:
To determine the efficacy of decitabine followed by Rapamycin in previously untreated elderly patients not able to receive standard chemotherapy or in patients with relapsed or refractory AML, through measurement of Complete Remission (CR), Complete Remission Incomplete Platelet Recovery (CRp), Partial Remission (PR), and event free and overall survival (Arm A).

To determine the safety of administration of decitabine with escalating doses of Ribavirin in elderly leukemia patients or patients with relapsed/refractory disease with M4/M5 subtypes anticipated to express high eukaryotic translation initiation factor 4E (eIF4E) at diagnosis (Arm B).

To establish effect of these sequential treatments on expression of phosphoinositide 3-kinase/protein kinase B/mammalian target of rapamycin (PI3K/Akt /mTOR) pathway proteins and on eukaryotic translation initiation factor 4E (eIF4E) activation through Western blot and phospho-flow methodologies.

To correlate the clinical response with baseline expression of phospho-p70S6 Kinase/phosphorylated protein kinase B (pAKT) and with the in vitro inhibitory effects of mammalian target of rapamycin (mTOR) inhibition with rapamycin or ribavirin on the level of downstream effectors.

To determine whether a leukemia stem cell phenotype is inhibited by the sequential administration of decitabine/rapamycin or decitabine/ribavirin.

ELIGIBILITY:
Inclusion Criteria:

4.1.1 Age >/= 18 4.1.2 Diagnosis of AML according to World Health Organization (WHO) criteria except acute promyelocytic leukemia AND 4.1.3 Refractory AML defined as failure to achieve Complete Remission (CR) after 2 cycles of induction chemotherapy or persistence of > 40% bone marrow blasts after one cycle of chemotherapy induction OR 4.1.4 Relapsed AML defined as any evidence of disease recurrence after achieving a documented first or greater Complete Remission (CR) OR 4.1.5 Relapsed AML after stem cell transplantation. 90 days (since stem cell infusion) must have elapsed between transplant and emergence of recurrent AML OR 4.1.6 Newly diagnosed AML in a patient >65 years old not considered fit for standard 7+ 3 chemotherapy or who declines such therapy after discussion of therapeutic options available.

4.1.7 Eastern Cooperative Oncology Group (ECOG) performance status <3

Exclusion Criteria:

4.2.1 Abnormal renal function as evidenced by a calculated creatinine clearance ≤ 30 ml/min (Cockcroft-Gault formula (Appendix 2) 4.2.2 Abnormal liver function: Bilirubin >2.0 mg/dl, transaminase(s) more than 2.5x the upper limits of normal 4.2.3 Active systemic infection not responding to antibiotics 4.2.4 Known diagnosis of human immunodeficiency virus infection (HIV) 4.2.5 Patients who are post-allogeneic transplantation should not have active Graft vs. Host Disease (GVHD) greater than grade 1 of skin at time of enrollment. They may have had donor lymphocyte infusion (DLI) but not within 4 weeks of beginning the study.

4.2.6 Pregnant or breastfeeding female subjects 4.2.7 Known or suspected Central Nervous System (CNS) leukemia involvement; past involvement is not an exclusion.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Liesveld, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Liesveld JL, Baran A, Azadniv M, Misch H, Nedrow K, Becker M, Loh KP, O'Dwyer KM, Mendler JH. A phase II study of sequential decitabine and rapamycin in acute myelogenous leukemia. Leuk Res. 2022 Jan;112:106749. doi: 10.1016/j.leukres.2021.106749. Epub 2021 Nov 11. PMID 34839054

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 37 patients signed consent for the study and 27 patients enrolled. Reasons for non-enrollment were withdrawal of consent (3 patients), diagnosis of MDS vs. AML on screening marrow (2 patients), enrollment on an alternate clinical trial (4 patients), and expiration during screening period due to sepsis (1 patient). The first patient enrolled in March 2014 and the last in January 2020.
Groups:
- Decitabine Followed by Rapamycin: Decitabine 20 mg/M2/day will be given as an IV infusion daily for 10 consecutive days starting on day 1 of cycle 1; in subsequent cycles, decitabine will be given for five days (days 1-5). Rapamycin 6mg (loading dose) will be administered on day 6; thereafter 2 mg/day on days 11-22 in cycle 1 and on days 6-22 in subsequent cycles. (Arm A: for patients with non-morphologic M4/M5 subtypes).
  Decitabine
- Decitabine Followed by Ribavirin: Decitabine 20 mg/M2/day will be given as an IV infusion daily for 10 consecutive days starting on day 1 of cycle 1; in subsequent cycles, decitabine will be given for five days (days 1-5). Ribavirin will be dosed from day 11-day 28 beginning with dose level 1 (1000mg orally twice daily). Number of patients with Dose Limiting Toxicities (DLT) at a given dose level is 0 of out of 3: enter 3 patients at the next dose level (dose Level 2- 1200mg orally twice daily; and then dose Level 3-1400 mg orally twice daily).(Arm B: For patients with morphologic M4/M5 subtypes).
  Decitabine
Period: Overall Study
Arm/Group | Decitabine Followed by Rapamycin | Decitabine Followed by Ribavirin
Started | 26 | 1
Completed | 24 | 0
Not Completed | 2 | 1
Not completed — Death | 1 | 1
Not completed — no marrow exam | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decitabine Followed by Rapamycin | Decitabine Followed by Ribavirin | Total
Number analyzed (Participants) | 26 | 1 | 27
Age, Continuous [Median (Full Range); unit: years] | 74 [31 to 86] | 80 [80 to 80] | 74 [31 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 0 | 15
  Male | 11 | 1 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 25 | 0 | 25
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 23 | 0 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 26 | 1 | 27

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival
Time Frame: 2 years
Population: The Ribavirin arm did not complete the study and entered hospice before 4 weeks. Median survival of the rapamycin arm included all 26 participant who started the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Decitabine Followed by Rapamycin | Decitabine Followed by Ribavirin
Number analyzed (Participants) | 26 | 0
months | 6.9 [4.8 to 12.2] |

2. Secondary Outcome: Blast Percentage in Peripheral Blood
Description: bone marrow aspirate and biopsy exam
Time Frame: baseline and four weeks
Population: Data was not collected for two patients in the rapamycin arm and 1 patient in the ribavirin arm.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Decitabine Followed by Rapamycin | Decitabine Followed by Ribavirin
Number analyzed (Participants) | 24 | 0
percentage of cells
  baseline | 24.7 (5.9) |
  week 4 | 14.7 (5.6) |

3. Secondary Outcome: Mean Change in Blast Percentage in Marrow
Description: Complete blood count with differential.
Time Frame: baseline and four weeks
Population: Data was not collected for two patients in the rapamycin arm and 1 patient in the ribavirin arm.
Measure: Mean (Full Range); unit: percentage of cells
Arm/Group | Decitabine Followed by Rapamycin | Decitabine Followed by Ribavirin
Number analyzed (Participants) | 24 | 0
percentage of cells | -18.5 [-86 to 64] |

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Decitabine Followed by Rapamycin | Decitabine Followed by Ribavirin
All-Cause Mortality (participants affected / at risk) | 25/26 | 1/1
Serious Adverse Events (participants affected / at risk) | 21/26 | 1/1
Other Adverse Events (participants affected / at risk) | 26/26 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine Followed by Rapamycin (N=26) | Decitabine Followed by Ribavirin (N=1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
pneumonia (Infections and infestations) | 0 | 1
syncope (Nervous system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 11 | 0
Intracranial hemorrhage (Nervous system disorders) | 3 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
decreased platelet count (Blood and lymphatic system disorders) | 1 | 0
skin infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Chest pain (General disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine Followed by Rapamycin (N=26) | Decitabine Followed by Ribavirin (N=1)
alkaline phosphatase increased (Hepatobiliary disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Confusion (Psychiatric disorders) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Hallucinations (Psychiatric disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 0
Infection (Infections and infestations) | 2 | 0
Lethargy (Nervous system disorders) | 2 | 0
Peripheral Neuropathy (Nervous system disorders) | 2 | 0
Presyncope (Nervous system disorders) | 2 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rhinitis/sinusitis (Infections and infestations) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0
Thromboembolic event (Vascular disorders) | 2 | 0
Fatigue (General disorders) | 16 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 | 0
Nausea (Gastrointestinal disorders) | 10 | 0
Constipation (Gastrointestinal disorders) | 9 | 0
Edema (General disorders) | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Headache (Nervous system disorders) | 6 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 0
Fever (General disorders) | 5 | 0
Hypotension (Vascular disorders) | 5 | 1
Skin infection (Infections and infestations) | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Bruising (Injury, poisoning and procedural complications) | 4 | 0
Chills (General disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
GI discomfort (Gastrointestinal disorders) | 4 | 0
Oral pain (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
ALT increased (Hepatobiliary disorders) | 3 | 0
Anxiety (Nervous system disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Dizziness (Nervous system disorders) | 3 | 0
Bleeding from central line (Blood and lymphatic system disorders) | 3 | 0
Extremity pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Hemorrhoids (Gastrointestinal disorders) | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0
Malaise (General disorders) | 3 | 0
Sore throat (Gastrointestinal disorders) | 3 | 0
Decreased platelets (Blood and lymphatic system disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Sepsis (Immune system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT02109744/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT02109744/ICF_001.pdf